CLINICAL TRIAL: NCT00559013
Title: Peri-Strips Dry With Veritas Collagen Matrix Staple Line Reinforcement for Colorectal Surgery
Brief Title: Peri-Strips Dry (PSD) Veritas Collagen Matrix Staple Line Reinforcement for Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CP1011, Rev C
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Results first posted 2012-05-24 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
Keywords: Staple line reinforcement; Staple line buttress; Anastomotic reinforcement
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): PSD Veritas Collagen Matrix Reinforcement Arm
  Interventions: Device: Staple line reinforcement

INTERVENTIONS:
Device: Staple line reinforcement — Placement of reinforcement material on circular anastomotic staple line for prevention of leak during and post surgery.

SUMMARY:
Purpose of the study is to assess the utility of PSD Veritas as a staple line reinforcement to minimize the risk of leakage during or after colo-rectal surgery.

DETAILED DESCRIPTION:
Study is designed as a prospective enrollment of patients undergoing open or laparoscopic colorectal surgery requiring the creation of an anastomosis. Patients who are scheduled for elective resection of the left, anterior and low anterior colon can be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must comply with follow-up evaluations
* Patient or representative must provide informed consent prior to enrollment
* Patient scheduled for elective surgical excision of the left, anterior or low anterior colon
* Patient must meet all criteria and be eligible to have open or laparoscopic colorectal surgery with primary anastomosis at one location

Exclusion Criteria:

* Crohns disease
* Emergency colorectal surgery for trauma, obstruction, ischemic bowel, perforated diverticulum and all other emergent diagnosis.
* Patients who have not had mechanical bowel preparation
* Patients with known documented sensitivity/allergy to bovine material
* Severe radiation damage to tissue
* Carcinomatosis or stage IV cancer
* BMI is 35 or greater
* Cancer at primary anastomosis site that cannot be excised
* Patients who require an ileo rectal anastomosis
* Surgery anticipated to include jejunostomy pouch
* Anticipated diverting stoma
* No anti adhesive barrier can be used around anastomotic site
* No multiple circular anastomosis
* Surgeons discretion to exclude any patient he/she feels would not have a safe anastomosis
* Patient life expectacny less than follow-up timeframe of study
* Pregnancy
* Patients currently enrolled in a study that competes for the same patient population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Karulf, MD, Principal Investigator — Colon & Rectal Surgery Associates
Locations (2):
- United States (2):
  - Lahey Clinic, Burlington, Massachusetts
  - Colon & Rectal Surgery Associates, Saint Paul, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 subjects were recruited from two principal investigators and their respective surgical hospitals in the US from approximately February 2007 through October 2008.
Pre-assignment Details: Subjects were excluded from the study if the met any of the exclusion criteria including having a a body mass index greater than 35, a history of Chron's Disease, or stage IV cancer. There was no washout, run-in or transition period to this study.
Groups:
- PSD Veritas Collagen Matrix Reinforcement Arm: Subjects receiving PSD Veritas Collagen Matrix for staple line reinforcement when undergoing open or laparoscopic colorectal surgery requiring the creation of an anastomosis.
Period: Overall Study
Arm/Group | PSD Veritas Collagen Matrix Reinforcement Arm
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PSD Veritas Collagen Matrix Reinforcement Arm
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.26 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Colorectal Related Adverse Events: Leak, Stricture and Hemorrhage.
Time Frame: Discharge and 1 Month post surgery
Measure: Number; unit: Participants
Arm/Group | PSD Veritas Collagen Matrix Reinforcement Arm
Number analyzed (Participants) | 38
Participants | 4

ADVERSE EVENTS:
Arm/Group | PSD Veritas Collagen Matrix Reinforcement Arm
Serious Adverse Events (participants affected / at risk) | 3/38
Other Adverse Events (participants affected / at risk) | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSD Veritas Collagen Matrix Reinforcement Arm (N=38)
Anastomotic Buttress Leak (Surgical and medical procedures) | 3 (3)
Bleeding (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSD Veritas Collagen Matrix Reinforcement Arm (N=38)
Post operative ileus (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No